CLINICAL TRIAL: NCT01532674
Title: Clinical, Microbiological and Biochemical Effects of the Antimicrobial Photodynamic Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Francisco Alpiste Illueca (Other)
Collaborators: Ondine Research Laboratories (Industry); Spanish Society of Periodontology and Osseointegration ( SEPA) (Unknown)
Responsible Party: Sponsor-Investigator, Francisco Alpiste Illueca, University Professor of University of Valencia, University of Valencia
Organization: University of Valencia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UV1
Record Dates: First submitted 2011-11-09; First posted 2012-02-14 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Root Planing; Tooth Exfoliation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antimicrobial photodynamic therapy (Experimental): Antimicrobial photodynamic therapy and scaling and root planing
  Interventions: Device: Antimicrobial photodynamic therapy (Periowave) and scaling and root planing
- scaling and root planing (Active Comparator): Only scaling and root planing
  Interventions: Procedure: scaling and root planing

INTERVENTIONS:
Device: Antimicrobial photodynamic therapy (Periowave) and scaling and root planing — ROOT PLANNING PROCEDURE:
  The procedure is the same as in the control group
  APPLICATION PROCEDURES OF THE PHOTOSENSITIZING AGENT :
  The photosensitive agent : Formulation Periowave Treatment Kit-2ml
  * Application of the photosensitive using a blunt needle at the bottom of the periodontal pocket with circular movements covering the entire perimeter of the tooth.
  * Application of diode laser with a peak of 8.5 cm. long with a curvature of 60 degrees and flexible. Making a move in and out from the apical region to the more coronal region of the periodontal pocket. Each tooth has a working time of 60 seconds.
  * All the periodontal pockets will be treated subgingivally
  * Elimination of the photosensitive by irrigation
  Other Names: Periowave
  Arms: Antimicrobial photodynamic therapy
Procedure: scaling and root planing — ROOT PLANNING PROCEDURE:
  An unique operator ( independent from the explorer) will do the root planing for both the test and control group.
  Every procedure will be done under local anaesthesia: Ultracain with Epinephrine 40/0,01 mg/ml. NORMON. It will be done a first session of root planning in the first and forth quadrant and in a 48 hours the root planning of the second and the third quadrant will be done. Every session wil be done with this material: Ultrasonic: Satelec suprasson p5 with ultrasonic tip H3, manual scalers: HU-FRIEDY 1/2, 7/8, 11/12, 13/14, 13/14 columbia.
  * The session will finish as soon as the operator have removed all the supragingival and subgingival calculus and plaque.
  Arms: scaling and root planing

SUMMARY:
The goal of this study is to determine if patients with chronic periodontitis when undergoing with scaling and root planing (SRP) plus photodynamic therapy in comparison with SRP alone result in improved clinical, microbiological and biochemical outcomes.

DETAILED DESCRIPTION:
This research is orientated to find an effective way to kill oral microorganisms that cause periodontitis and gingivitis with no problems of resistance, as it happens when we use antibiotics. The efficacy of this low power laser has been demonstrated in numerous fields in medicine and have been use it for years. The application of the photodynamic therapy is easy since we only have to fill the periodontal pocket with the photosensitive agent and apply the low power laser in that area. The photosensitive agent stain the bacteria immediately and the laser disrupts its membrane by a free-radical reaction. Improving the health status of the patients in a few weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic generalized moderate-advanced periodontitis: based on "Classification System for Periodontal Diseases and Conditions" Armitage 1999. (24).Extension of the 30 % of affected zones. Severity base on clinical attachment loss: moderate = 3-4 mm of CAL, severe= > or equal 5 mm CAL.
2. The subject is diagnosed with moderate or advanced chronic periodontitis.
3. The subject has at least 4 sites with PD of ≥5 mm + bleeding in at least two quadrants of the mouth.
4. A signed Informed Consent will be obtained.
5. The subject is an adult male or female > 18 years of age.
6. The subject has >18 fully erupted teeth, at least 3 teeth in each quadrant with one or more posterior teeth per quadrant (3º molars excluded).
7. The subject is willing and able to return for treatment and evaluation procedures scheduled throughout the course of this clinical study.

Exclusion Criteria:

1. The subject is pregnant or nursing or plans to become pregnant in the next 6 months.
2. The subject is a current smoker.
3. The subject has an active malignancy of any type by subject report.
4. The subject has chronic disease or diminished mental capacity that would mitigate the ability to comply with the protocol.
5. The subject has any significant chronic disease (either acute or chronic) or who is taking a medication with concomitant oral manifestations that in the opinion of the investigator would interfere with evaluation of safety or efficacy of the study.
6. The subject has an active periapical abscess or periodontal abscess or a history of acute necrotizing ulcerative gingivitis.
7. The subject has been treated with antibiotics within the 3-month period prior to beginning the study or any systemic condition which requires antibiotic coverage for routine periodontal procedures (e.g. heart conditions, joint replacements, etc.) by report of the subject.
8. The subject has a known allergy to Methylene Blue, polimetil metacrilate or chlorhexidine.
9. The subject Has severe glucose-6-phosphate dehydrogenase (G6PD) deficiency by subject report.
10. The subject currently uses anti-coagulant therapy at therapeutic doses.
11. The subject is currently using any photosensitizing medications.
12. Patients who have received SRP or Periodontal supportive therapy in the last 6 months
13. It is considered > 30% of plaque of an index of 2 or more in the Silness y Löe plaque index the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Improvement in Clinical Attachment Level | 6 months

SECONDARY OUTCOMES:
Improvement in Periodontal Pocket Depth | 6 months
Improvement in Bleeding on Probing | 6 months
Levels of IL-1 | 6 months.
levels of IL-6 | 6 months
Levels of FNT-alfa | 6 months
Levels of RANKL-OPJ. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alpiste Illueca Francisco, Professor, Principal Investigator — University of Valencia; Segarra vidal marta, postgraduate, Study Director — University of Valencia; López Roldán Andrés, Professor, Study Chair — University of Valencia; Puchades Rufino Juan, professor, Study Chair — University of Valencia; gil loscos francisco, professor, Study Chair — University of Valencia
Locations (1):
- University of Valencia, Valencia, Valencia, Spain